CLINICAL TRIAL: NCT03860337
Title: The Effect of Alginate on Carbohydrate and Fat Digestion in a Mixed Meal - A Pilot Trial
Brief Title: The Effect of Alginate on Carbohydrate and Fat Digestion in a Mixed Meal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Newcastle University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: SAU 01615
Record Dates: First submitted 2019-02-28; First posted 2019-03-01 (Actual); Last update posted 2019-10-02 (Actual); Status verified 2019-09

CONDITIONS: Triacylglycerol Digestion
Keywords: fat digestion; alginate; sausages

STUDY DESIGN:
Intervention Model Description: Double blind randomised controlled trial
Who Masked: Participant, Investigator
Masking Description: neither the researcher or the participant will know if the participant is eating alginate or control sausages
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alginate then Control (Experimental): This group will be given the alginate then the control sausages
  Interventions: Dietary Supplement: Alginate Sausage; Other: Control Sausage
- Control then Alginate (Experimental): This group will be given the control then alginate sausages
  Interventions: Dietary Supplement: Alginate Sausage; Other: Control Sausage

INTERVENTIONS:
Dietary Supplement: Alginate Sausage — Alginate sausage
Other: Control Sausage — Control Sausage

SUMMARY:
This study will investigate the effect of an extract of brown seaweed, called alginate, on fat digestion. The extract has been cooked into sausages and the alginate sausages will be compared to the same sausages that do not contain alginate. People taking part in the study will come to the study centre twice. Once to have the alginate sausage meal or the normal sausage meal and on the second visit they will have the other meal so then end up having had both types of sausages. The level of fat in their blood will be monitored over the four hours after the meal. The rate and amount of fat that moves into the blood after a meal is an indication of the amount of fat digestion. We believe that less fat will be digested and move into the blood when the volunteers eat the alginate sausages compared to the normal sausages.

DETAILED DESCRIPTION:
Alginate is an extract of brown seaweed and has been shown to reduce lipase activity in vitro. Lipase is a valid target for anti-obesity products as shown by the pharmaceutical drug orlistat which targets the same enzyme. Reducing the amount of lipase activity will reduce the amount of triacylglycerol (TAG) that will be digested and therefore absorbed and will be seen as a reduction in the level of circulating TAG in the blood. Adding alginate to a range of food products that are simple to include into the diet could help with the management of obesity. In this study, sausages containing alginate have been manufactured for us along with matched control sausage. The circulating TAG in the blood will be measured via fingerpick blood samples every 30 minutes for four hours after the volunteers have eaten either alginate sausages or normal sausages. The volunteers will come for two visits and consume the other sausage meal at the second so they will have had both types of sausage.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* pregnant or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-05-13 (Actual); Primary Completion 2019-06-19 (Actual); Study Completion 2019-06-19 (Actual)

PRIMARY OUTCOMES:
Concentration of circulating TAG in blood | 4 hours after the test meal
  mmol/L

SECONDARY OUTCOMES:
Concentration of circulating glucose in blood | 4 hours after the test meal
  mmol/L

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey P Pearson, PhD, Principal Investigator — Newcastle University
Locations (1):
- Newcastle University, Newcastle, Tyne and Wear, United Kingdom